CLINICAL TRIAL: NCT00089804
Title: A Randomized, Double-Blind, Placebo-Controlled, Three-Arm, Parallel-Group, Multicenter, Multinational Safety and Efficacy Trial of 300 mg and 900 mg of Abetimus Sodium in Systemic Lupus Erythematosus (SLE) Patients With a History of Renal Disease
Brief Title: Study of LJP 394 in Lupus Patients With History of Renal Disease
Acronym: ASPEN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim efficacy analysis indicated it would be futile to continue study.
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Michael J. Tansey, Chief Medical Officer, La Jolla Pharmaceutical Company
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LJP 394-90-14
Record Dates: First submitted 2004-08-13; First posted 2004-08-17 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Nephritis
Keywords: Lupus; Nephritis; Kidney; SLE; Systemic Lupus Erythematosus; Nephritis, Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Nephritis | interventions — abetimus; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 300 mg (three 2 mL vials of abetimus sodium plus six 2 mL vials of normal saline) administered i.v (in the vien) weekly
  Interventions: Drug: abetimus sodium (LJP 394) and/or placebo solution
- 2 (Active Comparator): 900 mg (nine 2 mL vials of abetimus sodium) administered i.v. (in the vein) weekly
  Interventions: Drug: abetimus sodium (LJP 394)
- 3 (Placebo Comparator): A volume of 18 mL (Nine 2 mL vials) of identically appearing placebo (phosphate-buffered saline) administered i.v. (in the vien) weekly
  Interventions: Drug: Phosphate-buffered saline

INTERVENTIONS:
Drug: abetimus sodium (LJP 394) and/or placebo solution — 300 mg (50 mg/mL)abetimus sodium (three 2 mL vials of of abetimus sodium plus six 2 mL vials of normal saline) administered i.v. (in the vien) weekly for 52 weeks
  Arms: 1
Drug: abetimus sodium (LJP 394) — 900 mg (50 mg/mL) abetimus sodium (nine 2 mL vials) administered i.v. (in the vien) weekly for 52 weeks.
  Arms: 2
Drug: Phosphate-buffered saline — A volume of 18 mL (nine 2 mL vials of normal saline) of identically appearing placebo (phosphate-buffered saline) administered i.v. (in the vien) weekly for 52 weeks
  Other Names: Placebo, normal saline
  Arms: 3

SUMMARY:
The primary purpose of this study is to determine whether abetimus sodium is more effective than placebo in delaying time to renal flare in SLE patients with a history of renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Lupus Erythematosus (SLE)
* Active SLE renal disease within past 4 years.
* Males or females between 12 and 70 years old.
* Females must be non-pregnant and non-lactating. Females and males must use adequate birth control methods during course of study.
* Ability to have weekly intravenous (IV) administration of study treatment.

Exclusion Criteria:

* Active SLE renal disease within past 3 months prior to entering study.
* Use of the following therapies within 3 months prior to entering the study: alkylating agents, e.g., cyclophosphamide, TNF inhibitors, cyclosporine.
* Use of mycophenolate mofetil that exceeds 1000 mg/day, azathioprine that exceeds 100 mg/day, methotrexate that exceeds 10 mg/week, leflunomide that exceeds 10 mg/day within 2 months prior to entering study.
* Use of rituximab within 6 months prior to entering study.
* Current abuse of drugs or alcohol.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 943 (Actual)
Dates: Start 2004-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To determine whether abetimus sodium is more effective than placebo in delaying the time to renal flare in SLE patients with a history of SLE renal disease. Weekly administration with a 52-week treatment duration. | Time to event (12 months fixed treatment duration)

SECONDARY OUTCOMES:
To determine whether treatment with abetimus sodium is more effective than placebo in delaying the time to Major SLE flare; and to determine whether treatment with abetimus sodium (LJP 394) is more effective than placebo in reducing proteinuria. | 12 month fixed treatment duration

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Tansey, MD, Ph.D., Study Director — Chief Medical Officer, La Jolla Pharmaceutical Company
Locations (201):
- United States (32):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Wallace Rheumatic Study Center, Los Angeles, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Private Practice, San Mateo, California
  - CRIA Research, Fort Lauderdale, Florida
  - Miami Children's Hospital, Miami, Florida
  - Emory University School of Medicine, Renal Division, Atlanta, Georgia
  - Private Practice, Augusta, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - Intermountain Orthopedics, Boise, Idaho
  - Rheumatology Associates, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - SOMARC Trials, LLC, Greenbelt, Maryland
  - Nephrology Associates, PC, Flushing, New York
  - North Shore - LIJ Health System, Lake Success, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - Seligman Center for Advanced Therapeutics, NYU Hospital for Joint Diseases, New York, New York
  - AAIR Research Center, Rochester, New York
  - Suny Upstate Medical University, Syracuse, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Private Practice, Camp Hill, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Arthritis Clinic, 371 North Parkway, Suite 400, Jackson, Tennessee
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Miracle Medical Clinic, 1170 Blalock Road, Houston, Texas
  - Renal Care Clinic, P.A., 17202 Red Oak Drive, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - San Antonio Kidney Disease Center, San Antonio, Texas
  - Clinical Research & Consulting Center, Fairfax, Virginia
  - Arthritis Northwest PLLC, Spokane, Washington
- Argentina (8):
  - CIR Hospital Sirio Libanes. Campana 4658, Buenos Aires, Ciudad Autonma de
  - Instituto CAICI, Rosario, Santa Fe Province
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Organización Médica de la Investigación, Buenos Aires, Uruguay 725 P.B.
  - Unidad de Alergia, Asma e Inmunología Clínica, Buenos Aires
  - Centro de Investigaciones en Enfermedades Reumaticas (CIER), Buenos Aires
  - Centro de Investigaciones Reumatologicas y Osteologicas, Buenos Aires
  - Investigación Clínica Polivalente, La Plata
- Australia (3):
  - Rheumatology Clinic, Cairns
  - Dept Medicine, Level 3 Wallace Freeborn Building, Royal North Shore Hospital, Pacific Highway, St Leonards
  - Vincents Hospital Daly Building, 41 Victoria Parade Fitzroy, Victoria
- Belarus (6):
  - Gomel Regional Clinical Hospital, Homyel
  - Minsk City Clinical Hospital # 2, Minsk
  - Minsk City Clinical Hospital # 164, Minsk
  - Minsk City Clinical Hospital # 9, Minsk
  - Minsk Regional Clinical Hospital, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Brazil (14):
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul-PUCRS, Porto Alegre-RS, Av. Ipiranga, 6690-Conj. 220-Jardim Botanico
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro, Avenida 28 de Setembro, 77
  - Hospital Hehopolis, São Paulo, Avenida Almirante Delamare, 1534-Sacoman
  - Hospital Geral de Goiania, GO Av Anhanguera 6479 Setor Oeste, Goiania-GO, Goiás
  - Santa Casa de Misericórdia de BeloHorizonte, Av. Francisco Sales, n. 1111 9 andar Ala D/ CCIH, Belo Horizonte, Minas Gerais
  - Hospital das Clinicas da Faculdade de Medicina da Universidade, Federal de Goiás, Servico de Reumatologia / 2 andar, Goiänia, Goiás, Primeira Avenida S/n Setor Universitário
  - Hospital e Maternidade Celso Pierro - PUCCampinas, Av. John Boyd Dunlop, s/n, Campinas - Sāo Paulo
  - Hospital de Clinicas - Universidade Estadual de Campinas - UNICAMP, Rua Vital Brasil, 250 - 3º andar - Cidade Universitária Zeferin, Campinas - SP
  - Athritis Clinica de Doenças Reumaticas, Av. Padre Anchieta, 1846 cj 1108, Curitiba - PR
  - Hospital de Clinicas de Porto Alegre - HCPA, Porto Alegre-RS
  - Hospital das Clínicas of Medicine School of University of São Paulo (USP) at Ribeirão Preto Rheumatology Department Avenida dos, Ribeirão Preto
  - Hospital Santa Izabel, Praca Almeida Couto, 500 - Naxaré, Salvador - BA
  - Irmandade da Santa Casa de Misericórdia de Sāo Paulo Rua, Dr. Cesário Motta Junior, 112, São Paulo
  - Rua Pedro de Toledo 1800 9 andar/ Ala central - Diretoria de Servico de Reumatologia, Săo Paulo - SP
- Bulgaria (6):
  - NMTranspH "Tsar Boris Treti", Clinic of Internal Diseases, Sofia, 104 "Maria Louisa" Blvd.
  - MHAT "Stara Zagora", Second Clinic of Internal Diseases, Stara Zagora, 11 "Armeiska" Street
  - MHAT "Sveti Ivan Rilski", Clinic of Rheumatology, Sofia, 13 "Urvich" Street
  - MHAT "Sveti Georgi", Clinic of Rheumatology, Plovdiv, 15A "Vasil Aprilov" Blvd.
  - Military Medical Academy, Clinic of Urology and Nephrology, Sofia, 3, Georgi Sofiiski, Str.
  - Clinic of Nephrology, MHAT "Alexandrovska" 1, Georgi Sofiiski, str.,, Sofia
- Czechia (3):
  - Fakultni nemocnice Plzen, Oddeleni klinické farmakologie, Pilsen, Edvarda Benese
  - VFN Prahal Lékarská fakulta, Klinika detského a dorostového lékarstvi,, Prague, Ke Karlovu, 09 Praha 2,
  - Revmatologický ústav, Prague
- Academic VL Tsitlanadze Scientific - Practical Center of Rheumatology, Tbilisi, Georgia
- Germany (5):
  - Herz and Rheumazentrum Kerckhoff-klinik GmbH, Bad Nauheim, Benekestrasse 2-8
  - Charité-Unversitätmedizin Berlin, CharitéCentrum Inn ere Medizin und Dermatologie, Berlin, Chariteplatz 1
  - Medizinische Klinik und Poliklinik IV des Universitätsklinikum Lepizig, Rheumatologie, Leipzig, Liebigstrasse 22
  - Georg August Universität Göttingen Universitätsklinikum, Zentrum Innere Medizin, Göttingen, Robert-Kochstr. 40
  - Johannes Gutenberg-Universität I. Medizinische Klinik und Poliklinik,Langenbeckstr. 1, Mainz
- Hong Kong (2):
  - Hong Kong University, Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
- Hungary (5):
  - Szent Margit Hospital, Department of Nephrology, Budapest
  - Diagnostic Units Hungary Kft., Budapest
  - Szent László Kórház, VI. Fertőző Belosztály, Budapest
  - Debrecen Medical University, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Immunnephrologia es Hypertonia Osztaly, Győr
- India (30):
  - Global Hospitals, Hyderabaad, Andhra Pradesh
  - Department of Nephrology, All India Institute of Medical Sciences, New Delhi, Ansari Nagar
  - Institute of Kidney Diseases and Research (IKRD) and Institute of Transplantation Sciences (ITS), Ahmedabad, Asarwa
  - Sri Ramachandra Medical College & Research Institute (Deemed University), Porur, Chennai
  - M.P. Shah Medical College & G.G. Hospital, Jamnagar, Gujarat
  - PVS Memorial Hospital Ltd., Kochi, Kaloor, Kerala
  - Apollo Gleneagles Hospital, Kolkata, Kankurgachi
  - St. Johns Medical College and Hospital, Dept. of Nephrology, Bangalore, Karnataka
  - M.S. Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Consultant and Head Department of Nephrology, Kamineni Hospitals, Hyderabaad, L.B. Nagar
  - Apollo Specialty Hospitals, Lake View Road, K.K., Nagar, Madurai, Tamil Nadu
  - Fortis Hospital, Dept. of Nephrology & Hypertension, Noida, Uttar Pradesh
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Devaki Hospital Ltd., Dept. of Nephrology, Chennai
  - Madras Institute of Nephrology, Vijaya Health Center, Chennai
  - Spectra Apollo Research Foundation, Chennai
  - Medwin Hospital, Hyderabaad
  - Nizams Institute of Medical Sciences, Hyderabaad
  - Department of Nephrology, CARE Hospital, Banjara Hills, Hyderabad
  - Armenian Church Trauma Center - Unit of Rabindranath Tagore International Institute of Cardiac Sciences, Kolkata
  - Sanjay Ghandi Post Graduate Institute of Medical Sciences, Lucknow
  - BYL Nair Charitable Hospital & TN Medical College, Mumbai
  - Seth G.S. Medical College & KEM Hospital, Mumbai
  - P.D. Hinduja National Hospital and Research Center, Mumbai
  - Department of Nephrology, JSS Hospital, Ramanuja Road, Mysore
  - Indraprastha Apollo Hospital, New Delhi
  - Jehangir Hospital, 32 Sassoon Road, Pune
  - Medical College Trivandrum, Trivandrum
  - King George Hospital, Visakhapatnam
- Indonesia (3):
  - Dept. of Internal Medicine, Saiful Anwar General Hospital, Malang, Jl. J.A. Suprapto No. 2
  - RS Kramat 128, Jakarta, Jl. Kramat Raya, Pusat
  - RS Hasan Sadikin, Bandung, Jl. Pasir Kaliki No. 190, Jawa Barat
- Italy (3):
  - Arcispedale S. Anna, Divisione di Reumatologia, Ferrara, Corso Giovecca 203
  - Azienda Ospedaliera Cattedra di Reumatologia, Padua, Via Giustiniani, 2
  - Universita di Pisa, Dipartimento di Medicina Interna, Pisa, Via Roma 67
- Lebanon (5):
  - Rayak Hospital, Riyaq, Bekaa Valley
  - Albert Haykel Hospital, Haykaliyeh-Tripoli
  - Nabatieh Governmental Hospital, Nabatieh
  - Hammoud Hospital University Medical Center, Saida
  - Labib Medical Center, Saida
- Malaysia (3):
  - Department of Medicine, Hospital Pulau Pinang,, Pulau Pinang, Jalan Residensi
  - CAPD Unit, Queen Elizabeth Hospital,, Sabak Bernam, Kota Kinabalu
  - Department of Medicine, Sarawak General Hospital, Jalan Tun Ahmad Zaidi Adruce,, Sarawak, Kuching
- Mexico (10):
  - Instituto Nacional de Ciencias Medicas y Nutricion "Salvador Zubiran", Departmento de inmunologia y Reumatologia, Delagacion Tlalpan, D.F.
  - Clínica de Diagnóstico y Tratamiento de las Enfermedades Reumáticas, Mexico City, D.F.
  - Blvd. Sanchez Taboada 9250-28 - Private Practice, Tijuana, Estado de Baja California
  - Hospital Aranda de la Parra, León, Guanajuato
  - Colomos #2292, Col. Providencia, Guadalajara, Jalisco
  - Centro de Estudios de Investigación Básica y Clínica S.C., Guadalajara, Jalisco
  - Hospital Star Medica, Morelia, Michoacán
  - Poliplaza Medica, Chihuahua City
  - Reumatologia, Mexicali
  - Hospital Privado San José de Ciudad Obregón, S.A. de C.V. Coahuila No. 263 Sur. Col. Centro. Ciudad Obregón, Sonora
- Philippines (4):
  - Chung Hua Hospital, Cebu
  - Davao Doctors Hospital, Davao City
  - Philippine General Hospital, Manila
  - Joint and Bone Center, University of Santo Tomas Hospital, Manila
- Poland (8):
  - Klinika Medycyny, Transplantacyjnej i Nefrologii in Warszawa, Nowogrodzka 59, At SPZOZ Szpital Kliniczny, Warsaw, Dzieciatka Jezus-Centrum Leczenia Obrażeń, Lindleya 4
  - Klinika Nefrologii, Transplantologii i Chorob Wewnetrznych - Akademickie Centrum Kliniczne - Szpital AMG, Gdansk
  - Klinika Chorob Wewnetrznych i Reumatologii - Gornoslaskie Centrum Medyczne, SPSK Nr 7 SL A M, Katowice
  - Oddzial Kiliniczny Nefrologii Hipertensjologii i Transplantologii Nerek SPZOZ, Uniwersytecki Szpital Kliniczny nr 1, Lodz
  - Klinika Reumatologii i Ukladowych Chorob Tkanki Lacznej, Lublin
  - Akademii Medycznej w Poznaniu, Zaklad Reumatologii i Immunologii Klinicznej, Poznan
  - Klinika Chorób Tkanki Łącznej, Warsaw
  - Klinika Nefrologii Dializoterapii I Chorob Wewnetrznych - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Portugal (5):
  - Centro Hospitalar de Lisboa Norte, EPE, Hospital de Santa Maria - Reumatologia, Lisbon, Av. Prof. Egas Moniz
  - Centro Hospitalar do Porto, EPE - Hospital de Santo Antonio, Departamento de Medicina - Unidade de Imunologia Clinica, Porto, Largo Prof. Abel Salazar
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia, Rua Conceicao Fernandes
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital de Egas Moniz, Unidade de Reumatologia, Lisbon, Rua Da Junqueira, 126
  - Hospital de Sāo Jeāo, Servico de Nefrologia, Porto
- RCMI Clinical Research Center, 1st Floor University Hospital Medical Center, San Juan, Puerto Rico
- Romania (4):
  - "Sf. Maria" Clinical Hospital, Bucharest
  - "Ion Stoia" Center of Rheumatic Diseases, Bucharest
  - Emergency Clinical County Hospital Cluj, Cluj-Napoca
  - Rehabilitation Clinical Hospital, Iași
- Serbia (4):
  - Institute of Nephrology and Urology Clinical Centre of Serbia, Belgrade
  - Institute of Rheumatology, Belgrade
  - University Medical Centre "Zvezdara", Clinical Department for Renal Diseases, Dimitrija Tucovica 161, Belgrade
  - Institute of Prevention, Treatment and Rehabilitation of Rheumatoid and Cardiovascular Patients "Niska Banja", Niška Banja
- Slovakia (2):
  - Reumatologicka ambulancia Fakultna nemocnica F D Roosevelta, Banska, Bystrica
  - Reumatologicka ambulancia Fakultna nemocnica s poliklinikou Milosrdni bratia spol s r o, Bratislava
- South Korea (9):
  - Ewha Woman's University College of Medicine, Mockdong Hospital, Seoul, Yangcheon-Gu
  - Inha University Hospital, Incheon
  - Bundang Cha General Hospital, Pochon Cha University, Kyonggi-do
  - Pusan National University Hospital, Pusan
  - Seoul National University Hospital, Department of Internal Medicine, Seoul
  - The Hospital for Rheumatic Disease, Hanyang University Medical Center, Seoul
  - Kangnam St. Mary's Hospital, Catholic University of Korea, Seoul
  - St. Mary's Hospital, Catholic University of Korea, Seoul
  - Ajou University Medical Center, Ajou University School of Medicine, Suwon
- Spain (3):
  - Hospital Clinic i Provincial de Barcelona, Centre Ciutat, Facultat de Medicina, Servicio de Enfermedades Autoinmunes, Barcelona, Calle Villarroel, 170
  - Hospital Universitario La Paz, Servico de Medicine Interne Planta 10, Madrid, Paseo de La Castellana 261
  - Hospital Universitari Vall d'Hebron, Servicia Medicina Interna, Edificio General, 3a Planta, Barcelona, Paseo Valle de Hebron 119-129
- University Lupus Clinic of the Department of Clinical Medicine, Faculty of Medicine, University of Colombo, P.O. Box 271, No 25,, Colombo, Kynsey Road, Sri Lanka
- Taiwan (12):
  - Buddhist Dalin Tzu Chi General Hospital, Vice Superintendent Room, Dalin Town, Chia-Yi County
  - Kaohsiung University Medical Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Kaohsiung Hsien
  - Chang Gung Memorial Hospital - Keelung, Keelung
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Chang-Kung University Hospital, Tainan
  - Taipei Veterans General Hospital - Immunology & Rheumatology Office, Taipei
  - Chang Gung Memorial Hospital - Taipei, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
  - Chi Mei Foundation Hospital, Yongkang District
- Thailand (3):
  - Department of Medicine, King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital - Division of Allergy, Immunology & Rheumatology, Dept. of Medicine, Bangkok
  - Rheumatic Disease Unit, Department of Internal Medicine, Phramongkutklao Hospital and College of Medicine, Bangkok
- Ukraine (6):
  - Donetsk Central Municipal Clinical Hospital #1, Donetsk
  - Kyiv Central Municipal Clinical Hospital, Kyiv
  - M.D. Strazhesko Institute of Cardiology AMS Ukraine, Kyiv
  - Kyiv Regional Clinical Hospital, Kyiv
  - Lviv Municipal Public Clinical Hospital, Lviv
  - Vinnitsa Regional Clinical Hospital of MoH of Ukraine, Vinnitsa

REFERENCES:
- See also: Sponsor's website — http://www.ljpc.com